## The GlaxoSmithKline group of companies

208564

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for study 208564: |
|---|---|---|
| | | A phase 1, randomised, double-blind, placebo-controlled study of the safety, tolerability, pharmacokinetics and pharmacodynamics of single subcutaneous doses of GSK2330811 in healthy Japanese participants. |
| <b>Compound Number</b> | : | GSK2330811 |
| <b>Effective Date</b> | : | Refer to Document Date |

# **Description:**

- The purpose of the final RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 208564.
- This RAP will be provided to the study team members to convey the Statistical Analysis Complete (SAC) deliverables.

## Author(s):

| Authors | Date |
|-----------------------------------------------------------|-------------|
| PPD | 20 OCT 2020 |
| Statistician (Hep/GI Biostatistics) | 30-OCT-2020 |
| PPD | 01 DEC 2020 |
| Senior Statistician (Hep/GI Biostatistics) | 01-DEC-2020 |
| PPD | 20 NOV 2020 |
| Quantitative Clinical Pharmacology Director (Hep/GI CPMS) | 30-NOV-2020 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

208564

# **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|----------------------------------------------------------------|-------------|
| PPD | 02-DEC-2020 |
| Programming Manager (Hep/GI Clinical Programming) | |
| PPD | 01-DEC-2020 |
| Senior Director Clinical Development (Hep/GI and Fibrosis) | 01-DEC-2020 |
| PPD | 01-DEC-2020 |
| Global Clinical Development Manager | 01-DEC-2020 |
| PPD | 01-DEC-2020 |
| Clinical Development Director (Hep/GI and Fibrosis) | 01-DEC-2020 |
| PPD | 01-DEC-2020 |
| Clinical Data Manager | 01-DEC-2020 |
| PPD | |
| Senior Director Therapeutic Group, Global Regulatory & Quality | 02-DEC-2020 |

# Clinical Statistics and Clinical Programming Line Approvals: (Method: Veeva Clinical Vault eSignature)

| (1120mour + co+w chimieur + ware exignment) | |
|---|---|
| Approver | |
| PPD | |
| Director (Hep | o/GI Clinical Statistics) |
| (On behalf of | (Line Manager, Head – Statistics)) |
| PPD | |
| Manager (He | p/GI Clinical Programming) |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRODUCTION. | | 5 |
| 2. | SUMMARY OF KI | EY PROTOCOL INFORMATION | 5 |
| | | o the Protocol Defined Statistical Analysis Plan | |
| | | ective(s) and Endpoint(s) | |
| | | ign | |
| | | Analyses | |
| | | alyses | |
| | 2.6. Final Analy | yses | / |
| 3. | ANALYSIS POPU | LATIONS | 7 |
| | 3.1. Protocol D | eviations | 8 |
| 4. | | NS FOR DATA ANALYSES AND DATA HANDLING | 9 |
| | | atment & Sub-group Display Descriptors | |
| | | Definitions | |
| | | Derivations and Handling of Missing Baseline Data | |
| | | on of Covariates, Other Strata and Subgroups | |
| | | omparisons and Multiplicity | 10 |
| | | siderations for Data Analyses and Data Handling | 40 |
| | Convention | ns | 10 |
| 5. | | TION ANALYSES | |
| | 5.1. Overview | of Planned Study Population Analyses | 11 |
| 6. | EFFICACY ANAL | YSES | 11 |
| 7. | SAFETY ANALYS | SES | 12 |
| | 7.1. Adverse E | vents Analyses | 12 |
| | | boratory Analyses | |
| | 7.3. Other Safe | ety Analyses | 12 |
| 8. | IMMUNOGENICI7 | TY ANALYSES | 13 |
| _ | | | |
| 9. | | TIC ANALYSES Pharmacokinetic Analyses | |
| | | Endpoint / Variables | |
| | | 9.1.1.1. Drug Concentration Measures | |
| | | 9.1.1.2. Derived Pharmacokinetic Parameters | |
| | | Summary Measure | |
| | | Population of Interest | |
| | | Strategy for Intercurrent (Post-Randomization) Events | |
| 10. | PHARMACODYN | AMIC AND / OR BIOMARKER ANALYSES | 16 |
| | | y Pharmacodynamic (and / or Biomarker) Analyses | |
| | | Endpoint / Variables | |
| | | Summary Measure | |

208564

| | | 10.1.3.<br>10.1.4.<br>10.1.5. | Population of Interest | .16 |
|---|---|---|---|---|
| 11. | REFER | RENCES | | .18 |
| 12. | APPEN | NDICES | | .19 |
| | 12.1. | <b>Appendix</b> | 1: Schedule of Activities | .19 |
| | | 12.1.1. | Protocol Defined Schedule of Events | .19 |
| | 12.2. | <b>Appendix</b> | 2: Assessment Windows | .22 |
| | | 12.2.1. | Definitions of Assessment Windows for Analyses | .22 |
| | 12.3. | | 3: Study Phases and Treatment Emergent Adverse | |
| | | 12.3.1. | Study Phases | |
| | | 40.00 | 12.3.1.1. Study Phases for Concomitant Medication | |
| | 40.4 | | Treatment Emergent Flag for Adverse Events | |
| | 12.4. | | 4: Data Display Standards & Handling Conventions | |
| | | 12.4.1. | Reporting Process | |
| | | 12.4.2. | Reporting Standards for Pharmackingtic | |
| | | 12.4.3.<br>12.4.4. | Reporting Standards for Pharmacokinetic | |
| | 12.5. | . — | Reporting Standards for Target Engagement | .29 |
| | 12.5. | 12.5.1. | General | |
| | | 12.5.1. | Study Population | |
| | | 12.5.2. | Safety | |
| | 12.6. | | 6: Reporting Standards for Missing Data | |
| | 12.0. | 12.6.1. | Premature Withdrawals | |
| | | | Handling of Missing Data | |
| | | 12.0.2. | 12.6.2.1. Handling of Missing and Partial Dates | |
| | 12.7. | Appendix | 7: Values of Potential Clinical Importance | |
| | | | Laboratory Values. | |
| | | | ECG | |
| | | | Vital Signs | |
| | 12.8. | | 8: Abbreviations & Trademarks | |
| | | 12.8.1. | Abbreviations | .40 |
| | | 12.8.2. | Trademarks | .41 |
| | 12.9. | <b>Appendix</b> | 9: List of Data Displays | .42 |
| | | 12.9.1. | Data Display Numbering | .42 |
| | | 12.9.2. | Mock Example Shell Referencing | |
| | | 12.9.3. | Deliverables | |
| | | 12.9.4. | Study Population Tables | |
| | | 12.9.5. | Safety Tables | |
| | | 12.9.6. | Safety Figures | .48 |
| | | 12.9.7. | Pharmacokinetic Tables | |
| | | 12.9.8. | Pharmacokinetic Figures | |
| | | 12.9.9. | Pharmacodynamic (and / or Biomarker) Tables | |
| | | | Pharmacodynamic (and / or Biomarker) Figures | |
| | | | Pharmacokinetic / Pharmacodynamic Figures | |
| | | | ICH Listings | |
| | 10.10 | | Non-ICH Listings | |
| | 1Z. IU. | Appendix | 10: Example Mock Shells for Data Displays | . อฮ |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 208564:

| Revision Chronology: | | |
|----------------------|-------------|----------|
| 2019N406151_00 | 11-SEP-2019 | Original |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There was an unplanned interim analysis conducted due to safety related temporary study hold criterion being met and was not specified in the protocol.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the safety and tolerability of a single SC dose of GSK2330811 in healthy Japanese participants | <ul> <li>Number of participants reporting AEs.</li> <li>Number of participants reporting SAEs.</li> <li>Number of participants with vital signs (blood pressure, heart rate, body temperature) reaching a threshold of potential clinical importance</li> <li>Number of participants with treatment emergent abnormal ECG findings.</li> <li>Number of participants with CTCAE grade 1 or higher safety laboratory results (clinical chemistry, haematology values where CTCAE grading applies).</li> <li>Number of participants with treatment emergent abnormal urinalysis findings</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the pharmacokinetic (PK) profile of a single SC dose of GSK2330811 in healthy Japanese participants | Pharmacokinetic parameters (Cmax, AUC, CL/F, Tmax, t <sub>1/2</sub> , Vss/F) |
| To assess the potential for anti-drug<br>antibody formation following a single<br>SC dose of GSK2330811 in healthy<br>Japanese participants | Number of participants with anti-GSK2330811 antibodies |
| To assess effects of GSK2330811 on<br>platelets and haemoglobin in healthy<br>Japanese participants | <ul> <li>Platelet nadir</li> <li>Time to platelet nadir</li> <li>Haemoglobin nadir</li> <li>Time to haemoglobin nadir</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To explore the PD and the PK/PD relationship for GSK2330811 in the blood of healthy Japanese participants | <ul> <li>Serum levels of free OSM</li> <li>Serum levels of total OSM</li> <li>Levels of Thrombopoietin (TPO)</li> <li>Levels of Erythropoietin (EPO)</li> </ul> |

## 2.3. Study Design



# 2.4. Statistical Analyses

The primary objective of this study is to determine the safety and tolerability of single subcutaneous doses of GSK2330811 in healthy Japanese participants. No formal hypotheses are being tested in this study and therefore no statistical analysis is planned.

## 2.5. Interim Analyses

An unplanned unblinded review of available exposure time-course data from the ongoing study cohort was initiated due to a safety related temporary study hold criterion being met. The unblinded data provided to CPMS and analysis report was documented in trial master file.

# 2.6. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

### 3. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who signed the ICF and were screened for eligibility | <ul><li>Study Population</li><li>Screen Failures</li></ul> |
| Enrolled | All participants who signed the ICF and were randomized into the study. | Study Population |
| Safety | <ul> <li>All randomized participants who received a full dose of study treatment.</li> <li>Participants will be analysed according to the treatment they received.</li> </ul> | <ul><li>Study Population</li><li>Safety</li><li>PK/PD selected tables and figures</li></ul> |
| | Note: In the very unlikely case a participant is not<br>randomized but receives at least one dose of study<br>treatment, these participants will be listed separately. | |
| Pharmacokinetic<br>(PK) | All participants in the Safety population who received at least one active dose of study treatment and had at least 1 non-missing PK assessment (Non-quantifiable values will be considered as non-missing values). | <ul><li>PK</li><li>PK/PD selected figures</li></ul> |
| | Participants will be analysed according to the study treatment they received. | |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

208564

#### 3.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [Version 1, 25 Nov 2019].

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

A separate table and listing of all COVID-19 related protocol deviations will be provided to capture the impact on visits and assessments.

# 4. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 4.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | Reporting |
| Code | Description | Description | Order in TFL <sup>[1]</sup> |
| А | GSK2330811 450 mg <b>SC - PARALLEL</b> | GSK2330811 450 mg | 2 |
| Р | Placebo - PARALLEL | Placebo | 1 |

#### NOTES:

#### 4.2. Baseline Definitions

For all endpoints the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 (or Day -1 where applicable) assessments are assumed to be taken prior to first dose and used as baseline.

In case that triplicate assessments are performed, the mean of triplicate assessments at any given time point will be used as the value for that time point.

#### 4.2.1. Derivations and Handling of Missing Baseline Data

If baseline data is missing, no derivation will be performed, and baseline will be set to missing. The baseline definition will be footnoted on all change from baseline displays.

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit – Baseline) / Baseline] |
| Nadir | = Lowest post-baseline value of endpoint for a participant [1] |
| Time (Days) to Nadir | = Study Day of Nadir – 1 <sup>[1]</sup> |

#### NOTES:

- 1: When there are multiple instances of the lowest value then the nadir used for reporting will be the earliest occurrence of that value.
- Unless otherwise specified, the baseline definitions specified in Section 4.2. Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays. 'Note: Baseline is defined as the predose Day 1 assessment, unless unavailable, in which case it is the latest pre-dose assessment.'
- If there are multiple measurements (i.e. ECG) the derivation will be based on the average values where available.

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

208564

# 4.3. Examination of Covariates, Other Strata and Subgroups

There is no planned examination of covariates, other strata and subgroup analyses due to the small overall sample size.

# 4.4. Multiple Comparisons and Multiplicity

There is no adjustment for multiplicity in this phase 1 study.

# 4.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.2 | Appendix 2: Assessment Windows |
| 12.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 12.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 12.5 | Appendix 5: Derived and Transformed Data |
| 12.6 | Appendix 6: Reporting Standards for Missing Data |
| 12.7 | Appendix 7: Values of Potential Clinical Importance |

208564

## 5. STUDY POPULATION ANALYSES

# 5.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the 'Safety' population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

## 6. EFFICACY ANALYSES

There are no efficacy analyses included in this study.

### 7. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs) and Serious (SAEs) will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

# 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, haematology laboratory tests, urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 9: List of Data Displays.

Descriptive statistics (n, arithmetic mean, standard deviation, median, minimum, and maximum) will be calculated for nadirs for platelet count and haemoglobin.

Descriptive statistics (n, median, minimum, maximum and range) will also be calculated for time to nadir for platelet count and haemoglobin.

Laboratory safety will be graded using CTCAE criteria version 5. CTCAE grade 1 or higher safety laboratory results will be presented (where CTCAE grading applies).

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

A separate listing to capture the COVID-19 infection assessment of participants based on new eCRF page will be provided.

The details of the planned displays are presented in Appendix 9: List of Data Displays.

208564

# 8. IMMUNOGENICITY ANALYSES

The immunogenicity analyses will be based on the "Safety" population, unless otherwise specified. The immunogenicity analysis summarises the incidence of confirmed anti-drug antibodies and lists the titre of immunogenicity results.

Details of the planned displays are presented in Appendix 9: List of Data Displays.

### 9. PHARMACOKINETIC ANALYSES

# 9.1. Secondary Pharmacokinetic Analyses

## 9.1.1. Endpoint / Variables

#### 9.1.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 12.4.3 Reporting Standards for Pharmacokinetic).

#### 9.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed concentration. |
| | Determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax. |
| | Determined directly from the concentration-time data. |
| AUC(0-t) | • Area under the concentration-time curve from time zero to the time of last quantifiable concentration (C(t)). |
| | Calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-inf) | Area under the concentration-time curve from time zero to infinity |
| | <ul> <li>Calculated as AUC(0-inf)=AUC(0-t)+C(t)/lambda_z. AUC(0-inf) should not be reported if<br/>the area coming from extrapolation is greater than 20% of AUC(0-inf).</li> </ul> |
| %AUCex | The percentage of AUC (0-inf) obtained by extrapolation will be calculated as: |
| | [AUC(0-inf) – AUC(0-t)] / AUC(0-inf) x 100 |
| t1/2 | Terminal half-life |
| | Calculated as t1/2=ln2/lambda_z. |
| CL/F | Apparent systemic clearance |
| Vss/F | Apparent volume of distribution at steady state |
| tlast | Time of last quantifiable concentration |

#### NOTES:

- Additional parameters may be included as required.
- lambda\_z is the first order rate constant associated with the terminal (log-linear) portion of the curve. Estimated by linear regression of time vs. log concentration

## 9.1.2. Summary Measure

Descriptive statistics (n, arithmetic mean, standard deviation [SD], 95% CI, minimum, median and maximum) will be calculated for all PK concentrations over time and for the

derived PK parameters. In addition, for log-transformed PK parameter variables (i.e. Cmax, AUC(0-t), AUC(0-inf), CL/F, Vss/F, t1/2), geometric mean, 95% CI and %CV $_b$  will be provided. Plots of mean concentrations will also include standard deviation [SD] for the mean.

## 9.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

#### 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

A 'While on-study' strategy will be implemented for intercurrent events.

- Withdrawn participants may be replaced in the study. Replacement participants will be dosed with the planned treatment of the withdrawn participant.
- All available data from participants who were withdrawn from the study will be analysed and listed, and all available planned data will be included in summary tables and figures, unless otherwise specified.
- Non quantifiable data will be handled as per GUI 51487
- If anomalous concentration data is identified, the pharmacokineticist will:
  - o excludes the PK concentration data deemed to be anomalous
  - o documents the reason for exclusion in the 'Code' folder of the Phoenix Project
  - o communicates exclusion to Statistics and Programming

Note: Any exclusion of anomalous PK concentration data is documented in the clinical study report (CSR). Anomalous PK data is excluded from PK summaries and is flagged by asterisk or appropriate footnote in the PK data listings.

# 10. PHARMACODYNAMIC AND / OR BIOMARKER ANALYSES

# 10.1. Exploratory Pharmacodynamic (and / or Biomarker) Analyses

#### 10.1.1. Endpoint / Variables

| Parameter | Parameter description |
|-----------|------------------------------------------------------|
| Free OSM | Free OSM concentration in serum |
| Total OSM | Total OSM concentration in serum |
| TPO | Thrombopoietin concentration in serum |
| EPO | Erythropoietin concentration in platelet-poor plasma |

#### 10.1.2. Summary Measure

Descriptive statistics (n, arithmetic mean, standard deviation [SD], 95% CI, minimum, median and maximum) will be calculated for free and total OSM concentrations over time. Descriptive statistics (n. geometric mean and standard deviation [SD] on log scale, CVb%) will be calculated for log transformed total OSM concentration and ratio to baseline. Plots of individual, mean concentrations with SD and median concentrations with range for total OSM will be produced.

Total OSM parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Total OSM, Cmax, Tmax, AUC(0-t), AUC(0-inf), %AUCex, t1/2, CL/V, Vss/V, tlast might be calculated with non-compartmental analysis, from the serum concentration-time data, as data permits.

Only data listing provided for TPO and EPO concentrations.

#### 10.1.3. Population of Interest

The exploratory pharmacodynamics analyses will be based on the safety population, unless otherwise specified.

### 10.1.4. Strategy for Intercurrent (Post-Randomization) Events

A 'While on-study' strategy will be implemented for intercurrent events.

All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.

208564

# 10.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

208564

# 11. REFERENCES

GSK Document Number 2019N406151\_00. Study ID 208564: A phase 1, randomised, double-blind, placebo-controlled study of the safety, tolerability, pharmacokinetics and pharmacodynamics of single subcutaneous doses of GSK2330811 in healthy Japanese participants.11-SEP-2019.

# 12. APPENDICES

# 12.1. Appendix 1: Schedule of Activities

# 12.1.1. Protocol Defined Schedule of Events

# **Screening Period**

| Screening Procedure | Screening (up to 30 days prior to Day 1) |
|---|---|
| Informed Consent | X |
| Inclusion and Exclusion Criteria | X |
| Demography | X |
| Full Physical Exam (incl. weight and height) | X |
| Medical History and current medical conditions <sup>1</sup> | Х |
| Concomitant Medication Review | Х |
| 12 lead ECG in triplicate | Х |
| Vitals (blood pressure, heart rate, body temperature) <sup>2</sup> | Х |
| Breath Alcohol Screen | X |
| Urine Drug Screen | X |
| HIV, HBV and HCV Screen | Х |
| Tuberculosis (TB) Screening QuantiFERON | Х |
| Haematology/Clinical Chemistry/Urinalysis/Clotting | X |
| SAE Review | X |

<sup>1.</sup> To include substance usage, family history of premature cardiovascular disease, medication, drug/alcohol history

<sup>2.</sup> Vital signs are to be taken before blood collection for laboratory tests.

208564

# Treatment and Follow-Up Period

| Procedure | Day<br>-1 | | [ | Oay 1 | | | Day<br>2 | Day<br>3 | Day<br>5 | Day<br>7 | Day<br>10 | Day<br>14 | Day<br>21 | Day<br>28 | Day<br>42 | Day<br>56 | Day<br>84 | Day 126<br>(follow-up<br>visit)/Early<br>Withdrawal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | ±1<br>day | ±1<br>day | ±1<br>day | ±1<br>day | ±2<br>days | ±2<br>days | ±7<br>days | ±7 days |
| Admission | Х | | | | | | | | | | _ uu, | | _ uu, | | uuyo | uuyo | uuye | ±. uuye |
| In-patient Stay | Х | | | Χ | | | | | | | | | | | | | | |
| Discharge | | | | | | | Х | | | | | | | | | | | |
| Outpatient Visit | | | | | | | | Χ | Χ | Χ | Х | Х | Х | Χ | Χ | Х | Χ | Х |
| Inclusion and Exclusion Criteria | Х | | | | | | | | | | | | | | | | | |
| Breath Alcohol Screen | Х | | | | | | | | | | | | | | | | | |
| Urine Drug Screen | X | | | | | | | | | | | | | | | | | |
| | | Pre-<br>dose | 0h | 1h | 4h | 8h | 24h | | | | | | | | | | | |
| Dosing <sup>3</sup> | | | Х | | | | | | | | | | | | | | | |
| Injection Site Reaction Assessment | | X <sup>5</sup> | X <sup>5</sup> | | X5 | | X <sup>5</sup> | | | | | | | | | | | Х |
| Brief Physical Exam | Χ | | | | | | X <sup>1</sup> | | | | | | | | | | | |
| Full Physical Exam <sup>6</sup> | | | | | | | | | | | | | | | | | | Х |
| Haematology/Clinical Chemistry | Χ | X <sup>2</sup> | | | | | X <sup>1</sup> | Χ | Χ | Χ | Х | Х | X <sup>2</sup> | Х | Χ | Χ | Χ | Χ |
| Urinalysis | Χ | | | | | | | | | Х | | | Х | | | | Х | Χ |
| 12 lead ECG (triplicate) | | Х | | | | | | | | Х | | | Х | | | | Х | Χ |
| Vitals (blood pressure, heart rate, body temperature) <sup>4</sup> | Х | Х | | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X |
| PK Sampling | | Х | | | | X1 | X1 | Х | Χ | Х | Х | Х | Х | Х | Χ | Х | Χ | Χ |
| Free & Total OSM Sampling | | Х | | | | X1 | X1 | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Immunogenicity Sampling | | Х | | | | | | | | | | Х | | Х | | | | Х |
| TPO Sampling | | Х | | | | | | | Х | | Х | | Х | | | | Х | |
| EPO Sampling | | Х | | | | | | | | Х | | Х | Х | | | Х | | |
| Concomitant Medication Review | | | | | | | | Мо | nitored fro | om screei | ning until e | end of foll | ow-up vis | it | | | | |
| SAE/AE Review | | | | | | SAE | s collecte | ed from si | gning of c | consent fo | rm, AEs o | collected o | continuous | sly from ti | ne of dos | e | | |

208564

#### Footnotes:

- 1. All post dose time points are in reference to the first injection of IMP.
- 2. Day 1 Pre-dose sample and Day 21 sample will be fasted for approximately 12 hr and will include lipids
- 3. IMP administration consists of 3 syringes, all 3 syringes are to be administered as closely together in time as possible
- 4. Vital signs are to be taken before blood collection for laboratory tests.
- 5. Assessments should be conducted immediately before first injection (pre-dose) and immediately after last injection (0h). Post dose assessments (4h and 24h) to be conducted in reference to the last injection of IMP. Any injection site reactions to be captured through AE reporting.
- 6. Full physical exam at follow-up will not include height
- The timing and number of planned study assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments as the result of emerging pharmacokinetic/pharmacodynamic data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files but will not constitute a protocol amendment. The Competent Authority (CA) and ethics committee (EC) will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the informed consent form (ICF). The changes will be approved by the CA and the EC before implementation.

# 12.2. Appendix 2: Assessment Windows

For haematology, chemistry, vital signs, ECG, urinalysis, immunogenicity, PK and biomarker outputs (incl. summaries and figures), Unscheduled and early withdrawal assessments will be included (see Appendix 4: Data Display Standards & Handling Conventions and Appendix 9: List of Data Displays).

Where unscheduled and early withdrawal visits are included in outputs, the following visit slotting will apply. If more than one visit slots to the same analysis timepoint, the closest visit to the analysis timepoint will be included in the summary and figure.

# 12.2.1. Definitions of Assessment Windows for Analyses

| Analysis Set / Domain | Analys | is Window | Analysis Timepoint |
|---|---|---|---|
| | Beginning<br>Timepoint | Ending Timepoint | |
| Haematology and Chemistry | Days less than 0 | | Screening |
| | Day 1 | Day 1 | Day 1 |
| | Day 2 | Day 2 | Day 2 |
| | Day 3 | Day 4 | Day 3 |
| | Day 5 | Day 6 | Day 5 |
| | Day 7 | Day 8 | Day 7 |
| | Day 9 | Day 12 | Day 10 |
| | Day 13 | Day 17 | Day 14 |
| | Day 18 | Day 24 | Day 21 |
| | Day 25 | Day 34 | Day 28 |
| | Day 35 | Day 49 | Day 42 |
| | Day 50 | Day 63 | Day 56 |
| | Day 64 | Day 105 | Day 84 |
| | Day 106 | Day 133 | Day 126 |

| Analysis Set / Domain | Analys | Analysis Timepoint | |
|---|---|---|---|
| | Beginning<br>Timepoint | Ending Timepoint | |
| Vital signs | Days less than 0 | | Screening |
| | Day 1 - Pre dose | | Day 1 - Pre dose |
| | Day 1 - 1H | | Day 1 - 1H |
| | Day 1 - 4H | | Day 1 - 4H |
| | Day 1 - 8H | | Day 1 - 8H |
| | Day 2 | Day 2 | Day 2 |
| | Day 3 | Day 4 | Day 3 |
| | Day 5 | Day 6 | Day 5 |
| | Day 7 | Day 8 | Day 7 |
| | Day 9 | Day 12 | Day 10 |
| | Day 13 | Day 17 | Day 14 |

208564

| Analysis Set / Domain | Analys | Analysis Timepoint | |
|---|---|---|---|
| | Beginning<br>Timepoint | Ending Timepoint | |
| | Day 18 | Day 24 | Day 21 |
| | Day 25 | Day 34 | Day 28 |
| | Day 35 | Day 49 | Day 42 |
| | Day 50 | Day 63 | Day 56 |
| | Day 64 | Day 105 | Day 84 |
| | Day 106 | Day 133 | Day 126 |

| Analysis Set / Domain | Ana | Analysis Timepoint | |
|---|---|---|---|
| | Beginning<br>Timepoint | Ending Timepoint | |
| ECG and Urinalysis | Days less than 0 | | Screening |
| | Day 1 | Day 1 | Day 1 |
| | Day 2 | Day 14 | Day 7 |
| | Day 15 | Day 42 | Day 21 |
| | Day 43 | Day 105 | Day 84 |
| | Day 106 | Day 133 | Day 126 |

| Analysis Set / Domain | Analysis | Window | Analysis Timepoint |
|---|---|---|---|
| | Beginning Timepoint | Ending Timepoint | |
| PK/ Free and Total OSM | Day 1 - Pre dose | | Day 1 - Pre dose |
| | Day 1 - 8H | | Day 1 - 8H |
| | Day 2 | Day 2 | Day 2 |
| | Day 3 | Day 4 | Day 3 |
| | Day 5 | Day 6 | Day 5 |
| | Day 7 | Day 8 | Day 7 |
| | Day 9 | Day 12 | Day 10 |
| | Day 13 | Day 17 | Day 14 |
| | Day 18 | Day 24 | Day 21 |
| | Day 25 | Day 34 | Day 28 |
| | Day 35 | Day 49 | Day 42 |
| | Day 50 | Day 63 | Day 56 |
| | Day 64 | Day 105 | Day 84 |
| | Day 106 | Day 133 | Day 126 |

| Analysis Set / Domain | | Analysis | Analysis | |
|---|---|---|---|---|
| | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| Biomarker samples | EPO | Day 1 | Day 1 | Day 1 |
| (EPO/ TPO) | | Day 2 | Day 9 | Day 7 |

208564

| Analysis Set / Domain | | Analysis | Analysis | |
|---|---|---|---|---|
| | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| | | Day 10 | Day 17 | Day 14 |
| | | Day 18 | Day 34 | Day 21 |
| | | Day 35 | Day 133 | Day 56 |
| | TPO | Day 1 | Day 1 | Day 1 |
| | | Day 2 | Day 7 | Day 5 |
| | | Day 8 | Day 17 | Day 10 |
| | | Day 18 | Day 34 | Day 21 |
| | | Day 35 | Day 133 | Day 86 |

| Analysis Set / Domain | Analysis Window | | Analysis |
|---|---|---|---|
| | Beginning<br>Timepoint | Ending Timepoint | Timepoint |
| Immunogenicity | Day 1 | Day 1 | Day 1 |
| | Day 10 | Day 21 | Day 14 |
| | Day 22 | Day 56 | Day 28 |
| | Day 56 | Day 133 | Day 126 |

For PK and PD planned and unplanned assessments will be summarised and listed. PK NCA will use all available data and will use actual relative time, not planned relative time.

For all endpoints an early withdrawal assessment occurred at the time when a planned assessment for that endpoint would have occurred ( $\pm$  the visit window), the early withdrawal visit will be slotted to that planned assessment and included in summaries. Where the plots use time as the x-axis, the early withdrawal visit will be included regardless of when the data was collected relative to the study window. For log type data (i.e. AEs), all early withdrawal data will be included in summaries. All early withdrawal data will be listed.

208564

# 12.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 12.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date.

| Study Phase | Definition |
|-----------------------|----------------------------------------|
| Pre-Treatment | Date ≤ Study Treatment Start Date/Time |
| Treatment<br>Emergent | Date > Study Treatment Start Date/Time |

#### 12.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to study treatment |
| Concomitant | Any medication that is not a prior |

#### NOTES:

• Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 12.3.2. Treatment Emergent Flag for Adverse Events

Adverse Events will be flagged as Treatment Emergent as described in the table in Section 12.3.1, where the AE Start Date/Time will be considered.

# 12.4. Appendix 4: Data Display Standards & Handling Conventions

# 12.4.1. Reporting Process

| Software | | | |
|---|---|---|---|
| The currently supported versions of SAS software will be used. | | | |
| Reporting Area | Reporting Area | | |
| HARP Server | HARP Server : \\uk1salx00175.corpnet2.com | | |
| HARP Compound | Reporting effort (RE) name in RAP | Туре | HARP folder / RE name |
| | Unplanned IA | Interim analysis | internal_01,<br>internal_02 |
| | SAC | Pre-programming/<br>dry run | data_look_01,<br>data_look_02 |
| | SAC | Final | final_01 |
| <b>Analysis Datasets</b> | | | |
| - Analysis dataset | s will be erected according to | Integrated Data Standay | rde Library (IDCL) CCK ARD |

 Analysis datasets will be created according to Integrated Data Standards Library (IDSL) GSK A&R dataset standards.

#### **Generation of RTF Files**

RTF files will be generated for SAC

# 12.4.2. Reporting Standards

#### General

• The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- All data will be reported according to the actual treatment the participant received.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting
  of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
- Dates will be reported in the format DDMMMCCYY e.g. 01Jan2020 unless otherwise stated.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.

208564

- The impact of any major deviation from the planned assessment times and/or scheduled visit days
  on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be included in summary tables and figures. Assessment windows for the unscheduled and early withdrawal assessments are specified in Appendix 2: Assessment Windows.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| | N = the number of participants from the relevant analysis population for the group or subgroup. |
| | n = the number of participants counted for the summary statistic. |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 12.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| PC Windows Non-<br>Linear (WNL) File for<br>GSK2330811 | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487. Note: Concentration values will be imputed as per GUI_51487. Note: GSK2330811 concentration values will be imputed as per GUI_51487. |
| Pharmacokinetic Parameter Derivation | |
| PK Parameter to be Derived by Programmer | None |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to SOP_314000 If one or more non-quantifiable (NQ) values occur in a profile before the first measurable concentration, they will be assigned a value of zero concentration. For linear plots, zero concentration value(s) before the first measurable concentration will be included in the plot. For log-linear plots, zero concentration value(s) before the first measurable concentration will be assigned a missing value. If a single NQ value occurs between measurable concentrations in a profile, the NQ should generally be omitted (set to missing) in the derivation of pharmacokinetic parameters, statistical analysis, and the individual subject plots. If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual subject plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the |

208564

derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing).

NQs which occur after the last measurable concentration will be omitted (set to missing) in the derivation of pharmacokinetic parameters and from the individual subject plots. In some circumstances, there may be a pharmacokinetic rationale for fluctuation resulting in non-measurable concentrations in the middle of the concentration-time profile (e.g., entero-hepatic recycling, erratic absorption from transdermal/inhaled formulations). In these cases, the NQ values could be set to missing or to some other values (e.g., ½ LLQ) and subsequent valid concentrations may be retained. A reference line indicating LLQ will be included in plots.

For the calculation of mean or median pharmacokinetic profiles. When estimating the mean or median value for the concentration at a given time point (i.e., descriptive mean or median curve), the following guidelines should be considered:

All NQ values will be set to zero except when an individual NQ falls between two quantifiable values, in which case it will be omitted from the calculation of mean or median profiles. Measurable concentrations which follow more than one consecutive mid-profile NQ will be omitted (set to missing). The mean/median value at a time-point where one or more samples have NQ values will be reported (in tabular or graphical fashion) even if the mean/median value is below the LLQ of the assay. For linear plots, zero concentration value(s) will be included in the plot. For log-linear plots, zero concentration value(s) will be assigned a missing value.

Zero mean or median values will be included in summary tables. In certain cases, the NQ values could be set to missing or to some other values (e.g.,  $\frac{1}{2}$  LLQ) with proper scientific justification(s). A reference line indicating LLQ will be included in plots.

It should be noted that a high proportion of NQ values may affect the standard deviation (SD); if more than 30% of values are imputed, then SD will not be displayed. Any table of summary statistics for concentration-time data will report N (number of subjects in the analysis population), n (number of subjects with non-missing values) and number imputed (number of subjects with imputed values (i.e., NQ assigned zero concentration).

BQL (Below the Quantification Limit) may be displayed in listings by legacy systems instead of NQ; these abbreviations are interchangeable and mean that a sample has been received, analysed and a concentration below the LLQ of the assay found. Scientific judgement and prior knowledge should always be used in applying these guidelines.

Descriptive Summary Statistics, Graphical Displays and Listings Refer to IDSL PK Display Standards.

Refer to GUI 51487

208564

# 12.4.4. Reporting Standards for Target Engagement

| Total OSM Concentra | ition Data |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| PC Windows Non-<br>Linear (WNL) File for<br>Total OSM | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487. Note: Total OSM concentration values will be imputed as per GUI_51487. |
| Total OSM Parameter | Derivation |
| Total OSM Parameter to be Derived by Programmer | None |
| Total OSM Parameter | Data |
| Is NQ impacted Total OSM Parameters Rule Being Followed | Yes, refer to SOP_314000. If one or more non-quantifiable (NQ) values occur in a profile before the first measurable concentration, they will be assigned a value of zero concentration. For linear plots, zero concentration value(s) before the first measurable concentration will be included in the plot. For log-linear plots, zero concentration value(s) before the first measurable concentration will be assigned a missing value. If a single NQ value occurs between measurable concentrations in a profile, the NQ should generally be omitted (set to missing) in the derivation of total OSM parameters, statistical analysis, and the individual subject plots. If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual subject plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of total OSM parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing). NQs which occur after the last measurable concentration will be omitted (set to missing) in the derivation of pharmacokinetic parameters and from the individual subject plots. For the calculation of mean or median total OSM profiles. When estimating the mean or median value for the concentration at a given time point (i.e., descriptive mean or median value for the concentration at a given time point (i.e., descriptive mean or median curve), the following guidelines should be considered: All NQ values will be set to zero except when an individual NQ falls between two quantifiable values, in which case it will be omitted from the calculation of mean or median profiles. Measurable concentrations which follow more than one consecutive mid-profile NQ will be omitted (set to missing). The mean/median value at a time-point where one or more samples have NQ values will be reported (in tabular or graphical fashion) even if the mea |

208564

| | Any table of summary statistics for concentration-time data will report N (number of subjects in the analysis population), n (number of subjects with non-missing values) and number imputed (number of subjects with imputed values (i.e., NQ assigned zero concentration). BQL (Below the Quantification Limit) may be displayed in listings by legacy systems instead of NQ; these abbreviations are interchangeable and mean that a sample has been received, analysed and a concentration below the LLQ of the assay found. Scientific judgement and prior knowledge should always be used in applying these guidelines. |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to GUI_51487 |

## 12.5. Appendix 5: Derived and Transformed Data

#### 12.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Where multiple assessments are made, the mean of replicate assessments at any given time point will be used as the value for that time point. This derived mean will be reported in the listing in addition to the individual assessments.
- If there are two values within a time window, the value closest to the target day for that window will be
  used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Dose Date → Study Day = Ref Date Dose Date
  - Ref Data ≥ Dose Date → Study Day = Ref Date (Dose Date) + 1

## 12.5.2. Study Population

#### **Cumulative Dose**

Placebo: 0

GSK2330811: Number of Injections x 150

Dose unit: Milligram

## **Demographics**

### Age

- Only birth year is captured on the eCRF, therefore GSK standard ISDL algorithms will be used for calculating age where birth date will be imputed as follows:
- The missing date and month will be imputed as '30th June'
- Birth date will be presented in listings as 'YYYY'

#### **Body Mass Index (BMI)**

Calculated as Weight(kg)/Height(m)<sup>2</sup>

#### 12.5.3. Safety

#### **ECG Parameters**

#### **RR Interval**

If RR interval (msec) is not provided directly, then RR can be derived using machine read QTcF as:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

208564

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of decimal places in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 decimal places: '< x' becomes x 0.01
  - Example 2: 1 decimal places: '> x' becomes x + 0.1
  - $\circ$  Example 3: 0 decimal places: '< x' becomes x 1.

# 12.6. Appendix 6: Reporting Standards for Missing Data

# 12.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e. as specified in the protocol) was defined as completion of all assessment on Day 126. |
| | A maximum of 4 non-evaluable participants will be replaced. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed and<br/>all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Withdrawal visits will be slotted as per Appendix 2: Assessment Windows or will be summarised as withdrawal visits. |

# 12.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 12.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>In case of partial dates (i.e. day missing, only month and year present) recorded for AE start and end, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

208564

# 12.6.2.2. Imputation of Missing Data for OSM Free and Total

| Element | Reporting Detail |
|---|---|
| LLQ/2 | If data are missing due to readings being below the limits of quantification, then a value equivalent to LLQ/2 will be imputed. |
| | • If the readings are above the upper limit of quantification, the sample should be further diluted to be within the upper limit of quantification of the assay. The measured concentration should then be corrected for the additional dilution factor. |
| | These values will be used for the computation of the change from baseline and for summaries, plots and analysis, if deemed applicable. |
| | The number of data imputed will be highlighted in the summaries and figures, whereas listings will report the values as below LLQ. |
| | The numeric values and LLQ will be presented in listing as a reference, and the LLQ will be mentioned in footnotes where appropriate (e.g. figures). |

# 12.7. Appendix 7: Values of Potential Clinical Importance

# 12.7.1. Laboratory Values

Haematology and chemistry parameters will use CTCAE grades (CTCAE criteria, V5.0: November 27, 2017) to highlight important results based on laboratory value only (i.e. no clinical judgement will be applied). CTCAE grades will replace the category of "values of potential clinical importance" for haematology parameters, see table below for reference.

| Laboratory<br>Parameter | CTCAE<br>v5.0<br>Term for<br>Adverse<br>Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|
| Haemoglobin | Anemia | Hemoglobin<br>(Hgb) <lln<br>- 100 g/L</lln<br> | Hgb <100 -<br>80g/L | Hgb <80 g/L;<br>transfusion<br>indicated | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |
| Haemoglobin | Hemoglob in increased | Increase in >0 -<br>2 g/dL above<br>ULN or above<br>baseline if<br>baseline is<br>above ULN | Increase in<br>>2 - 4 g/dL<br>above ULN<br>or above<br>baseline if<br>baseline is<br>above ULN | Increase in >4<br>g/dL above ULN<br>or above<br>baseline if<br>baseline is<br>above ULN | - | - |
| Lymphocyte count | Lymphocy<br>te count<br>decrease<br>d | <lln -="" 0.8<br="">GI/L</lln> | <0.8 - 0.5<br>GI /L | <0.5 - 0.2<br>GI /L | <0.2 GI /L | - |
| Lymphocyte count | Lymphocy<br>te count<br>increased | - | >4 – 20<br>GI/L | >20 GI/L | - | - |
| Neutrophil count | Neutrophil<br>count<br>decrease<br>d | <lln -="" 1.5<br="">GI /L</lln> | <1.5 - 1.0<br>GI /L | <1.0 - 0.5<br>GI /L | <0.5 GI/L | - |
| Platelet count | Platelet count decrease d | <lln -="" 75.0="" gi<br="">/L</lln> | <75.0 - 50.0<br>GI /L | <50.0 - 25.0 GI | <25.0 GI/L | - |
| White blood cell count | Leukocyto sis | - | - | >100 GI/L | Clinical<br>manifestations<br>of leucostasis;<br>urgent<br>intervention<br>indicated | Death |
| White blood cell count | White blood cell | <lln -="" 3.0<br="">GI /L</lln> | <3.0 - 2.0<br>GI /L | <2.0 - 1.0<br>GI /L | <1.0 GI /L | - |

208564

| Laboratory<br>Parameter | CTCAE<br>v5.0<br>Term for<br>Adverse<br>Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|
| | decrease<br>d | | | | | |
| Alanine<br>Amino<br>Transferase<br>(IU/L) | Alanine<br>aminotran<br>sferase<br>increased | >ULN - 3.0 x<br>ULN if baseline<br>was normal; 1.5<br>- 3.0 x baseline<br>if baseline was<br>abnormal | >3.0 - 5.0 x<br>ULN if<br>baseline was<br>normal; >3.0<br>- 5.0 x<br>baseline if<br>baseline was<br>abnormal | >5.0 - 20.0 x<br>ULN if baseline<br>was normal;<br>>5.0 - 20.0 x<br>baseline if<br>baseline was<br>abnormal | >20.0 x ULN if<br>baseline was<br>normal; >20.0<br>x baseline if<br>baseline was<br>abnormal | |
| Aspartate<br>Amino<br>Transferase<br>(IU/L) | Aspartate<br>aminotran<br>sferase<br>increased | >ULN - 3.0 x<br>ULN if baseline<br>was normal; 1.5<br>- 3.0 x baseline<br>if baseline was<br>abnormal | >3.0 - 5.0 x<br>ULN if<br>baseline was<br>normal; >3.0<br>- 5.0 x<br>baseline if<br>baseline was<br>abnormal | >5.0 - 20.0 x<br>ULN if baseline<br>was normal;<br>>5.0 - 20.0 x<br>baseline if<br>baseline was<br>abnormal | >20.0 x ULN if<br>baseline was<br>normal; >20.0<br>x baseline if<br>baseline was<br>abnormal | |
| Calcium<br>(MMOL/L) | Hypocalc<br>emia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" <lln="" calcium="" l;="" l<="" lonized="" mmol="" td=""><td>Corrected serum calcium of &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;1.75 - 1.5 mmol/L; lonized calcium &lt;0.9 - 0.8 mmol/L; hospitalization indicated</td><td>Corrected serum calcium of; &lt;1.5 mmol/L; lonized calcium &lt;0.8 mmol/L; life-threatening consequences</td><td>Death</td></lln> | Corrected serum calcium of <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <1.75 - 1.5 mmol/L; lonized calcium <0.9 - 0.8 mmol/L; hospitalization indicated | Corrected serum calcium of; <1.5 mmol/L; lonized calcium <0.8 mmol/L; life-threatening consequences | Death |
| Cholesterol | Cholester ol - high | >ULN - 7.75<br>mmol/L | >7.75 -<br>10.34<br>mmol/L | >10.34 - 12.92<br>mmol/L | >12.92 mmol/L | |
| Creatinine | Creatinine increased | >ULN - 1.5 x<br>ULN | >1.5 - 3.0 x<br>baseline;<br>>1.5 - 3.0 x<br>ULN<br>Change in | >3.0 x baseline;<br>>3.0 - 6.0 x<br>ULN | >6.0 x ULN | |
| Glucose | Hyperglyc<br>emia | Abnormal glucose above baseline with no medical intervention | daily managemen t from baseline for a diabetic; oral antiglycemic agent initiated; | Insulin therapy initiated; hospitalization indicated | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>indicated | Death |
| Laboratory<br>Parameter | CTCAE<br>v5.0<br>Term for<br>Adverse<br>Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|
| | | | workup for diabetes | | | |
| | Hypoglyc | <lln -="" 3.0<br="">mmol/L</lln> | <3.0 - 2.2 | <2.2 - 1.7 | <1.7 mmol/L;<br>life threatening<br>consequences; | |
| Glucose | emia | | mmol/L | mmol/L | seizures | Death |
| Potassium | Hyperkale<br>mia | >ULN - 5.5<br>mmol/L | >5.5 - 6.0<br>mmol/L;<br>intervention<br>initiated | >6.0 - 7.0<br>mmol/L;<br>hospitalization<br>indicated | >7.0 mmol/L;<br>life-threatening<br>consequences | Death |
| | Hypokale | <lln -="" 3.0<="" td=""><td>Symptomatic with <lln -="" 3.0mmol="" indicated<="" intervention="" l;="" td=""><td>&lt;3.0 - 2.5<br/>mmol/L;<br/>hospitalization</td><td>&lt;2.5 mmol/L;</td><td></td></lln></td></lln> | Symptomatic with <lln -="" 3.0mmol="" indicated<="" intervention="" l;="" td=""><td>&lt;3.0 - 2.5<br/>mmol/L;<br/>hospitalization</td><td>&lt;2.5 mmol/L;</td><td></td></lln> | <3.0 - 2.5<br>mmol/L;<br>hospitalization | <2.5 mmol/L; | |
| Potassium | mia | mmol/L | | indicated | consequences | Death |
| Sodium | Hypernatr<br>emia | >ULN - 150<br>mmol/L | >150 - 155<br>mmol/L;<br>intervention<br>initiated | >155 - 160<br>mmol/L;<br>hospitalization<br>indicated | >160 mmol/L;<br>life-threatening<br>consequences | Death |
| Sodium | Hyponatre<br>mia | <lln -="" 130<br="">mmol/L</lln> | 125-129<br>mmol/L and<br>asymptomati<br>c | 125-129 mmol/L<br>symptomatic;<br>120-124 mmol/L<br>regardless of<br>symptoms | <120 mmol/L;<br>life-threatening<br>consequences | Death |
| Total | Blood<br>bilirubin | >ULN - 1.5 x<br>ULN if baseline<br>was normal; ><br>1.0 - 1.5 x<br>baseline if<br>baseline was | >1.5 - 3.0 x<br>ULN if<br>baseline was<br>normal; >1.5<br>- 3.0 x<br>baseline if<br>baseline was | >3.0 - 10.0 x<br>ULN if baseline<br>was normal;<br>>3.0 - 10.0 x<br>baseline if<br>baseline was | >10.0 x ULN if<br>baseline was<br>normal; >10.0<br>x baseline if<br>baseline was | |
| Bilirubin Triglycerides | hypertrigly ceridemia | abnormal 1.71 mmol/L - 3.42 mmol/L | abnormal<br>>3.42<br>mmol/L - 5.7<br>mmol/L | >5.7 mmol/L -<br>11.4 mmol/L | abnormal >11.4 mmol/L; life-threatening consequences | Death Death |

208564

## 12.7.2. Laboratory Values – Haematology, Chemistry and Liver

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Homotoorit | Ratio of 1 | Male | | 0.54 |
| Hematocrit | Rallo of 1 | $\Delta$ from BL | ↓0.075 | |
| Hamadahin | g/L | Male | | 180 |
| Hemoglobin | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umal/l | | | >1.3*ULN |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5x ULN |
| T. Bilirubin + ALT | µmol/L<br>U/L | High | 1.5x ULN T. Bilirubin<br>+<br>≥ 2x ULN ALT |

208564

## 12.7.3. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 12.7.4. Vital Signs

| Vital Sign Parameter Units | | Clinical Concern Range | |
|----------------------------|------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decr | ease | Incre | ease |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

208564

## 12.8. Appendix 8: Abbreviations & Trademarks

## 12.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AUC | Area Under the Curve |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CL/F | Apparent Clearance |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| LLN | Lower Limit of Normal |
| NCA | Non-Compartmental Analysis |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| tlast | Time of last quantifiable concentration |
| Tmax | Time of occurrence of Cmax |
| t1/2 | Half-life |
| ULN | Upper Limit of Normal |
| Vss/F | Steady state apparent volume of distribution |
| %AUCex | Percentage of AUC(0-inf) obtained by extrapolation |

208564

## 12.8.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
|---------------------------------------------------------|

None

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin

208564

## 12.9. Appendix 9: List of Data Displays

### 12.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|------------|
| Study Population | 1.1 to 1.11 | |
| Safety | 3.1 to 3.23 | 3.1 to 3.5 |
| Pharmacokinetic | 4.1 to 4.3 | 4.1 to 4.3 |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.6 | 6.1 to 6.3 |
| Pharmacokinetic / Pharmacodynamic | | 7.1 |
| Section | List | tings |
| ICH Listings | 1 to 27 | |
| Other Listings | 28 to 35 | |

## 12.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 12.9.3. Deliverables

| Delivery [1] | Description |
|--------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

208564

# 12.9.4. Study Population Tables

| Study I | Population Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition | Include total column | SAC |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| Protoc | ol Deviation | | | | - |
| 1.3. | Safety | DV1 | Summary of Important Protocol Deviations Not Related to COVID-19 | | SAC |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations Related to COVID-19 | | |
| Popula | tion Analysed | | | | |
| 1.5. | Screened | SP1 | Summary of Study Populations | | SAC |
| Demog | raphy | , | | 1 | , |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics | Include: Height, Weight, and BMI | SAC |
| 1.7. | Enrolled | DM11 | Summary of Age Ranges | | SAC |
| 1.8. | Safety | DM6 | Summary of Race and Racial Combinations | | SAC |
| Conco | mitant Medicati | ons and other Me | dical Conditions | | |
| 1.9. | Safety | MH4 | Summary of Past Medical Conditions | | SAC |
| 1.10. | Safety | MH4 | Summary of Current Medical Conditions | | SAC |
| 1.11. | Safety | CM8 | Summary of Concomitant Medications | | SAC |

208564

# 12.9.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.2. | Safety | AE5A | Summary of Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | SAC |
| 3.3. | Safety | AE1 | Summary of Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.4. | Safety | AE15 | Summary of Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 3.5. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 3.6. | Safety | AE3 | Summary of Serious Drug-Related Adverse Events by Overall Frequency | | SAC |
| 3.7. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | | SAC |
| Chemis | stry | | | | |
| 3.8. | Safety | LB1 | Summary of Chemistry | | SAC |
| 3.9. | Safety | LB17 | Summary of Worst-Case Chemistry Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.10. | Safety | SAFE_T1 | Summary of Chemistry Results by Maximum CTCAE Grade | Footnote: "CTCAE criteria, V5.0:<br>November 27, 2017" | SAC |
| Haemato | ology | • | | | <u>.</u> |
| 3.11. | Safety | LB1 | Summary of Haematology | By parameter | SAC |
| 3.12. | Safety | LB16 | Summary of Haematology Results by Maximum CTCAE Grade Increase Post-Baseline Relative to Baseline | Footnote: "CTCAE criteria, V5.0:<br>November 27, 2017" | SAC |
| 3.13. | Safety | LB17 | Summary of Worst Case Haematology Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | | SAC |
| 3.14. | Safety | SAFE_T2 | Summary of Nadirs for Selected Haematology Parameters | By parameter, treatment group Produce for Platelet count and Haemoglobin. Footnote: "Nadir is the lowest post- baseline value of the parameter" | SAC |
| 3.15. | Safety | SAFE_T3 | Summary of Days to Nadir of Selected Haematology<br>Parameters | by parameter, treatment group. Produce for Platelet count and Haemoglobin. Footnote: "Nadir is the lowest post- baseline value of the parameter" | SAC |

| Safety: 7 | Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Urinalys | is | | | | · |
| 3.16. | Safety | SAFE_T4 | Summary of Worst Case Urinalysis Results Post-Baseline Relative to Baseline | Tests to include: Urine blood, Urine Glucose (dipstick), Urine Ketones (dipstick), Urine Microscopy – Bacteria, Urine Microscopy - Red Blood Cells, Urine Microscopy - White Blood Cells, Urine Protein (dipstick), Urine Specific Gravity | SAC |
| ECG | | | | | |
| 3.17. | Safety | EG1 | Summary of ECG Findings | | SAC |
| 3.18. | Safety | EG2 | Summary of ECG Values | Footnote: Average used for triplicate ECG measurements | SAC |
| 3.19. | Safety | EG2 | Summary of Change from Baseline in ECG Values | Footnote: Average used for triplicate ECG measurements | SAC |
| Vital Sig | ns | | | | |
| 3.20. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC |
| 3.21. | Safety | VS7 | Summary of Worst Case Vital Signs Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | | SAC |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.22. | Safety | SAFE_T5 | Summary of Worst Case Vital Sign Results Relative to Change from Baseline Potential Clinical Importance (PCI) Criteria | | SAC |
| Immunog | enicity | | | | |
| 3.23. | Safety | IMM1 | Occurrence of Anti-Drug Antibodies | Add footnote: Note: The denominator for confirmed positive is the total number of subjects at that visit who have immunogenicity data available. | SAC |

#### 208564

# 12.9.6. Safety Figures

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Haema | atology | I | | | |
| 3.1. | Safety | SAFE_F1 | Subject Profiles for Haematology by Treatment Group | By Haematology parameter. This output should be produced for: Platelet Count, Haemoglobin Use rules for CTCAE boundaries X axis use 'Actual Relative Time (Days)' from dose. Show all observed values including unscheduled. Add footnote "Figure displays a subset of haematology parameters" Panel by treatment group | SAC |
| 3.2. | Safety | SAFE_F2 | Mean Profile for Haematology by Treatment Group | By Haematology parameter. This output should be produced for: Platelet Count, Haemoglobin X axis shows visits with approximate temporal spacing Add footnote "Figure displays a subset of haematology parameters" | SAC |
| 3.3. | Safety | SAFE_F3 | LFT Patient Profiles | ALT = Alanine Amino Transferase, AST = Aspartate Amino Transferase, Alk. Phos. = Alkaline Phosphatase, Total Bili. = Total Bilirubin | SAC |
| ECG | | | | | · |
| 3.4. | Safety | EG7 | Empirical Distribution Function for Maximum Change from baseline in QTcF Interval | Both treatments in one plot. Calculate maximum change from baseline. | SAC |

208564

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.5. | Safety | EG8 | Distribution of QTcF Change by Visit and Treatment | Use the 0, 30, 60 thresholds following shell. | SAC |

## 12.9.7. Pharmacokinetic Tables

| Pharma | cokinetic: Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | PK Concentration | | | | |
| 4.1. | PK | PKCT1 | Summary of Plasma GSK2330811 Concentration-Time Data | Note: LLQ=100 ng/mL. Values below LLQ have been imputed to 0. SD is set to missing if No. Imputed/n > 0.3. | SAC |
| Derived | I PK parameter | rs | | | |
| 4.2. | PK | PKPT1 | Summary of Derived Plasma Pharmacokinetic Parameters of GSK2330811 | | SAC |
| 4.3. | PK | PKPT3 | Summary of Log-Transformed Derived Plasma<br>Pharmacokinetic Parameters of GSK2330811 | | SAC |

208564

# 12.9.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | ncentration | | | | |
| 4.1. | PK | PKCF1P | Individual GSK2330811 Plasma Concentration-Time Plot by Subject (Linear and Semi-Log) | Footnote for all PK and PK/PD figures:<br>'LLQ is calculated at 100 ng/mL.<br>Values below LLQ have been imputed to 0.' Use actual time (days) as x axis<br>(where days is a continuous variable) | SAC |
| 4.2. | PK | PKCF4 | Mean (±SD) Plasma GSK2330811 Concentration-Time Plots by Treatment (Linear and Semi-log) | Use planned time (days) as x axis (where days is a continuous variable) | SAC |
| 4.3. | PK | PKCF5 | Median (Range) Plasma GSK2330811 Concentration-Time Plots by Treatment (Linear and Semi-log) | Use planned time (days) as x axis (where days is a continuous variable) | SAC |

#### 208564

# 12.9.9. Pharmacodynamic (and / or Biomarker) Tables

| Pharma | acodynamic (ar | nd or Biomarker): | Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serum | level of OSM | | | | |
| 6.1. | Safety | PD1 | Summary of Serum Level of Free OSM by Treatment Group | Calculate confidence intervals and add number imputed Add footnote: [1] No. of subjects with BLQs assigned half of the lower limit of quantification (LLQ = 2.5pg/ml) | SAC |
| 6.2. | Safety | PD1 | Summary of Serum Level of Total OSM by Treatment Group | Calculate confidence intervals and add number imputed Add footnote: [1] No. of subjects with BLQs assigned half of the lower limit of quantification (LLQ = 2.5pg/ml) | SAC |
| 6.3. | Safety | PD1 | Summary of Ratio of Serum Level of Total OSM to Baseline by Treatment Group | Calculate confidence intervals and add number imputed Add footnote: [1] No. of subjects with BLQs assigned half of the lower limit of quantification (LLQ = 2.5pg/ml) | SAC |
| 6.4. | Safety | PD2 | Summary of Log Transformed Serum Level of Total OSM by Treatment Group | Calculate confidence intervals and add number imputed Add footnote: [1] No. of subjects with BLQs assigned half of the lower limit of quantification (LLQ = 2.5pg/ml) | SAC |

| Pharmacodynamic (and or Biomarker): Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.5. | Safety | PKPT1 | Summary of Derived Serum Pharmacokinetic Parameters of Total OSM by Treatment Group | | SAC |
| 6.6. | Safety | РКРТ3 | Summary of Log-Transformed Derived Serum Pharmacokinetic Parameters of Total OSM by Treatment Group | | SAC |

#### 208564

# 12.9.10. Pharmacodynamic (and / or Biomarker) Figures

| riiaiiii | acodynamic (a | , | l iguico | 1 | T |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Serum | levels of OSM | <u> </u> | | | |
| 6.1. | Safety | PKCF1P | Individual Serum Level of Total OSM Concentration-Time Plot by Treatment (Linear and Semi-Log) | Add LLQ reference line Conditionally add ULQ reference line Page by treatment Total OSM: LLQ is calculated at 2.5pg/ml. Values below LLQ have been imputed to LLQ/2. Use actual time (days) as x axis (where days is a continuous variable) | SAC |
| | | | | Add Footnote to indicate amount of imputed data. | |
| 6.2. | Safety | PKCF4 | Mean (±SD) Serum Level of Total OSM Concentration-Time Plots by Treatment (Linear and Semi-log) | Add LLQ reference line Conditionally add ULQ reference line Use planned time (days) as x axis (where days is a continuous variable) Total OSM: LLQ is calculated at 2.5pg/ml. Values below LLQ have been imputed to LLQ/2. | SAC |
| 5.3. | Safety | PKCF5 | Median (Range) Serum Level of Total OSM Concentration-<br>Time Plots by Treatment (Linear and Semi-log) | Add LLQ reference line Conditionally add ULQ reference line Use planned time (days) as x axis (where days is a continuous variable) Total OSM: LLQ is calculated at 2.5pg/ml. Values below LLQ have been imputed to LLQ/2. | SAC |

208564

# 12.9.11. Pharmacokinetic / Pharmacodynamic Figures

| Pharmacokinetic / Pharmacodynamic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| OSM vs GSK23308 | 11 concentrat | ion | | | |
| 7.1. | PK | PKPD_F1 | Scatter Plot of Total Serum OSM vs Plasma Concentration of GSK2330811 | X axis: PK Page by visit Add LLQ reference lines for both Conditionally add ULQ reference line for total Footnotes: GSK2330811: LLQ is calculated at 100 ng/mL. Values below LLQ have been imputed to 0. Total OSM: LLQ is calculated at 2.5pg/ml. Values below LLQ have been imputed to LLQ/2. | SAC |

208564

# 12.9.12. ICH Listings

| ICH: Listin | ngs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject D | isposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | Enrolled | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | Enrolled | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | | SAC |
| 4. | Enrolled | TA1 | Listing of Planned and Actual Treatments | | SAC |
| Protocol [ | Deviations | | | | |
| 5. | Enrolled | DV2 | Listing of Important Protocol Deviations | | SAC |
| 6. | Enrolled | DV2 | Listing of COVID-19 related Protocol Deviations | | SAC |
| 7. | Enrolled | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Populatio | ns Analysed | | | | |
| 8. | Enrolled | SP3 | Listing of Subjects Excluded from Any Population | | SAC |
| Demograp | ohy | | | | |
| 9. | Enrolled | DM2 | Listing of Demographic Characteristics | | SAC |
| 10. | Enrolled | DM9 | Listing of Race | | SAC |
| Prior and | Concomitant Medic | ations | | | |
| 11. | Enrolled | CM3 | Listing of Concomitant Medications | | SAC |

| ICH: Listi | ngs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposure | and Treatment Cor | npliance | | | |
| 12. | Enrolled | EX3 | Listing of Exposure Data | Order by treatment, subject r. Include: Treamtent, Site ID/subjID, Start Datetime of Dose/Study day, Stop Datetime of Dose/Study day, Dose (this will be the cumulative dose) (eg450), Dose units, Root of administration, Number of injections | SAC |
| Adverse I | Events | | | | |
| 13. | Enrolled | AE8 | Listing of All Adverse Events | | SAC |
| 14. | Enrolled | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 15. | Enrolled | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Serious a | nd Other Significan | t Adverse Ever | nts | | |
| 16. | Enrolled | AE8CP | Listing of Serious Adverse Events | | SAC |
| 17. | Enrolled | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 18. | Enrolled | AE8CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |

| ngs | | | | |
|---|---|---|---|---|
| Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ogy | | | | |
| Enrolled | SAFE_L1 | Listing of All Haematology Values and Changes from Baseline | See listing 23 in 201246. Report:<br>Standard result, Change from<br>baseline and Percent change from<br>baseline. Do not flag CTCAE<br>grades | SAC |
| Enrolled | LB5 | Listing of Laboratory Values of CTCAE Grade | Include Haematology and clinical chemistry laboratory data | SAC |
| Enrolled | LB5 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | Include Haematology and clinical chemistry laboratory data | SAC |
| Enrolled | LB14 | Listing of Laboratory Data with Character Results | | SAC |
| | _ | | | |
| Enrolled | UR2 | Listing of Urinalysis Results | | SAC |
| Enrolled | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC |
| Enrolled | EG5 | Listing of Abnormal ECG Findings | | SAC |
| S | • | | | • |
| Enrolled | VS4 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | | SAC |
| enicity | | | | |
| Enrolled | IMM2 | Listing of Immunogenicity Results | | SAC |
| | Enrolled | Population IDSL / Example Shell DSL / Ex | Population Example Shell Title | Population Example Shell Title Programming Notes |

208564

# 12.9.13. Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK cor | PK concentration and derived PK parameters | | | | |
| 28. | PK | PKCL1 | Listing of GSK2330811 Plasma Concentration-Time Data | Add data dependent footnote: 'Note: NA=Not Available [data dependent], NQ=Non-Quantifiable, LLQ value=100ng/mL' | SAC |
| 29. | PK | PKCL1 | Listing of Derived GSK2330811 Pharmacokinetic Parameters | | SAC |
| Serum | levels of OSM | | | | |
| 30. | PK | PKCL1 | Listing of Serum Level of OSM | Include both Free and Total OSM Add footnote: 'Note: BLQ = Below the limit of quantification which is 2.5pg/ml for both free and total OSM' | SAC |
| 31. | Safety | PKCL1 | Listing of Derived Total OSM Pharmacokinetic Parameters | | SAC |
| Serum | levels of TPO | and EPO | | | |
| 32. | PK | PKCL1 | Listing of Level of Thrombopoietin in Serum | | SAC |
| 33. | PK | PKCL1 | Listing of level of Erythropoietin in Plasma | | SAC |
| Other | | | | | |
| 34. | Enrolled | PAN12 | Listing of COVID-19 Assessments and Symptom Assessments for Subjects with COVID-19 Adverse Events | | SAC |
| 35. | Enrolled | PAN7 | Listing of All Subjects with Visits and Assessments Impacted by COVID-19 Pandemic | | SAC |

208564

## 12.10. Appendix 10: Example Mock Shells for Data Displays

Example: SAFE\_T1
Protocol: 208564
Population: Safety


Test: Creatinine (UMOL/L)

Event: Creatinine increased

| Treatment | N | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|-------------------|----|---------|---------|---------|---------|
| Placebo | XX | XX | XX.X | XX.XX | XX.X |
| GSK2330811 450 mg | XX | XX | XX.X | XX.XX | XX.X |

Note: CTCAE criteria, V5.0: November 17, 2017 graded on laboratory test value.

Only events with at least one graded value are shown.

208564

Example: SAFE\_T2
Protocol: 208564

Protocol: 208564 Page 1 of n

Population: Safety

Table XX.XX

Summary of Nadirs for Selected Haematology Parameters [as Percent Change from Baseline]

| Lab Test (unit) | Treatment | N | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|
| Hemoglobin (G/L) | Placebo | XX | XX | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | GSK2330811 450 ma | XX | XX | XX.X | XX.XX | XX.X | XX.X | XX.X |

....

Note: Nadir is the lowest post-baseline value of the parameter.

208564

Example: SAFE\_T3
Protocol: 208564
Population: Safety


Table XX.XX

Summary of Days to Nadir for Selected Haematology Parameters

| Lab Test (unit) | Treatment | | n | Median | Min | Max | Range |
|------------------|-------------------|----|----|--------|-----|-----|-------|
| Hemoglobin (G/L) | Placebo | | XX | XX | XX | XX | XX |
| | GSK2330811 450 mg | XX | XX | XX | XX | XX | XX |

.....

Note: Nadir is the lowest post-baseline value of the parameter.

208564

Page 1 of 1

Example: SAFE T4

Programming note: please flag to study team/ statistics when summarizing if observe any character variables not the minimum value and not presented as an increase category.

Tests to summarise as X=BACTM URQ (minimum value=NONE SEEN)

Tests to summarise as Y= BLD\_URC, PROT\_URG, KETO\_URG, GLUC\_URG (minimum value=NEGATIVE)

Tests to summarise as Z= RBCM URG, WBCM URG (minimum value=NONE SEEN)

Tests to summarise as W= SG URG (minimum value=Low)

Example modified from UR1

Protocol: ABC123456
Population: Safety/Other study specific

| Test | - | Treatment A (N=248) | Treatment B (N=247) |
|------|---------------------|---------------------|---------------------|
| X | n | 230 | 232 |
| | No Change/Decreased | 222 (97%) | 223 (96%) |
| | Any Increase | 8 (3%) | 9 (4%) |
| | Increase to MANY | 6 (3%) | 5 (2%) |
| Y | n | 230 | 232 |
| | No Change/Decreased | 222 (96%) | 222 (96%) |
| | Any Increase | 7 (3%) | 10 (4%) |
| | Increase to TRACE | 2 (<1%) | 5 (2%) |
| | Increase to 1+ | 1 (<1%) | 4 (2%) |
| | Increase to 2+ | 1 (<1%) | 0 |
| | Increase to 3+ | 4 (2%) | 1 (<1%) |
| Z | n | 230 | 232 |
| | No Change/Decreased | 222 (96%) | 222 (96%) |
| | Any Increase | 7 (3%) | 10 (4%) |
| | Increase to 0-1 | 2 (<1%) | 5 (2%) |
| | Increase to 5-10 | 1 (<1%) | 4 (2%) |
| | Increase to 10-15 | 1 (<1%) | 0 |
| | Increase to 15-20 | 2 (<1%) | 1 (<1%) |

208564

| | Increase to 20-25<br>Increase to 25-50 | 2 (<1%)<br>4 (2%) | 0<br>1 (<1%) |
|---|---|---|---|
| W | n | 230 | 232 |
| | No Change/Decreased | 222 (97%) | 223 (96%) |
| | Any Increase | 8 (3%) | 9 (4%) |
| | Increase to NORMAL | 6 (3%) | 5 (2%) |
| | Increase to HIGH | 6 (3%) | 5 (2%) |

Note: Little n does not include Not done or No results.

208564

Example: SAFE\_T5
Protocol: 208564

Protocol: 208564 Page 1 of n

Population: Safety

| Test (Unit) | Change Category | Placebo<br>(N=XX) | GSK2330811 450 mg<br>(N=XX) |
|---|---|---|---|
| Diastolic blood pressure (mmHg) | n Decrease >= 10 Decrease >= 20 Increase >= 10 Increase >= 20 | xx<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) |
| Heart Rate (bmp) | n Decrease >= 15 Decrease >= 30 Increase >= 15 Increase >= 30 | xx<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx<br>xx (xx%)<br>xx (xx%) |
| Systolic blood pressure (mmHg) | n Decrease >= 20 Decrease >= 40 Increase >= 20 Increase >= 40 | xx (xx%) xx (xx%) xx (xx%) xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) |

208564

Example: SAFE\_F1
Protocol: 208564
Population: Safety


Figure XX.XX
Participant Profiles for Haematology by Treatment Group



Programming notes:

One legend including all participants.

Make plot as large as possible to fill space.

add (P) to denote placebo participants.

y-axis will be displayed on the left-hand side plot and the labels for the reference lines will be included on the right-hand side plot.

208564

Example: SAFE\_F2
Protocol: 208564
Population: Safety


Figure XX.XX Mean Profile for Haematology by Treatment Group



Programming notes:

See output 3.9 from 201247.

Make plot as large as possible to fill space.

Use different marker symbol, line pattern and colour by treatment group.

Table: Include N after treatment group and use same colour as in the plot.

208564

Example: SAFE\_F3
Protocol: 208564
Population: Safety


Figure XX.XX LTF Patient Profiles



Note: M = Male, F = Female, ALT = Alanine Amino Transferase, AST = Aspartate Amino Transferase, Alk. Phos. = Alkaline Phosphatase, Total Bili. = Total Bilirubin

Clinical Concern Levels: ALT, AST and Alk. Phos: 2 times respective ULN, Total Bili: 1.5 times the ULN

208564

Example: PKPD\_F1
Protocol: 208564
Population: PK


Figure XX.XX Scatter Plot of Free Serum OSM vs Plasma Concentration of GSK2330811



208564


Example: SAFE\_L1 Protocol: 208564

Population: Enrolled

Listing XX Listing of All Haematology Values and Changes from Baseline

| Lab Test<br>(Units) | Treatment | CentreID/<br>subjid | Visit/Analysis<br>visit | Date of collection | Study Day | Standard<br>Result | Change from<br>Baseline | Percentage<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| XX | | Xx/xx | XX | XX | XX | XX | XX | XX |

## Signature Page for 208564 TMF- 7927164 v 1.0

| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 07-Dec-2020 08:33:02 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 07-Dec-2020 14:00:17 GMT+0000 |

Signature Page for TMF-7927164 v1.0